CLINICAL TRIAL: NCT03489070
Title: A Randomized Controlled Trial to Compare the Efficacy of Traumastem® Versus Surgicel® for the Secondary Treatment of Local Bleeding in Patients Undergoing Hepatic Resection
Brief Title: Traumastem® Versus Surgicel® for the Secondary Treatment of Local Bleeding in Patients Undergoing Hepatic Resection
Acronym: TSFHR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jialin Zhang, Director of Hepatobiliary Surgery Department, Principal Investigator, Clinical Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Absorbable hemostatic gauze
Record Dates: First submitted 2018-03-24; First posted 2018-04-05 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Liver Hemorrhage
Keywords: Liver resection; Liver Hemorrhage; Traumastem; Surgicel
MeSH Terms: interventions — Surgicel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traumastem® (Active Comparator): Oxidized nonregenerated cellulose hemostatic agents.Traumastem® absorbable patches, applied topically, once, intraoperatively to stop bleeding.The patches are used on the wound surface of the liver.
  Interventions: Combination Product: Surgicel®
- Surgicel® (Active Comparator): Oxidized regenerated cellulose hemostatic agents.Surgicle® absorbable patches, applied topically, once, intraoperatively to stop bleeding.The patches are used on the wound surface of the liver.
  Interventions: Combination Product: Traumastem®

INTERVENTIONS:
Combination Product: Traumastem® — Intraoperative application as secondary hemostatic treatment
  Arms: Surgicel®
Combination Product: Surgicel® — Intraoperative application as secondary hemostatic treatment
  Arms: Traumastem®

SUMMARY:
Topical hemostats are agents that stop bleeding by contributing blood to clot. Oxidized cellulose, a sort of mechanical hemostatic material, predominantly forms a block to stop the blood flow and provides a surface to clot more rapidly.It was marketed for the first time in 1945 and widely used for its convenience, biocompatibility, and bactericide from that time. It is currently available in many commercial products, while manufactured using either a regenerated or nonregenerated process. The physicochemical property and hemostatic efficacy of oxidized regenerated cellulose (ORCG) and oxidized nonregenerated cellulose (ONRCG) has been well documented using in vitro test and animal models, and ONRCG was seemingly superior to ORCG in terms of hemostasis. However, no clinical study has been performed to verify. Therefore, the objective of this prospective randomized study is to assess the hemostatic efficacy of ORCG (Surgicel®, Ethicon) vs ONRCG (Traumastem®, Bioster) for hemostasis of local bleeding in patients undergoing hepatic resection.

DETAILED DESCRIPTION:
Representative liver resected surface (prominent bleeding site) was applied the ply of gauze with several seconds of even finger gentle press under aseptic conditions, then it was untouched and observed for 10 min. Vascular occlusion of the liver was allowed if necessary, but was open for evaluation of hemostatic efficacy. Hemostatic time began to calculate when gauze was applied. Time to hemostasis was recorded in seconds and the maximum time to hemostasis was 600 seconds. Hemostasis success was achieved based on there was no visible bleeding or minimal ooze from the resection wound.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with informed consent
* Adults aged between 18 to 75 and do not plan to have child within 1 year after the surgery
* Resection of at least the equivalent tissue volume of 1 anatomical segment of the liver
* Minor to moderate (oozing/diffuse) bleeding from the incisal area after conventional resection procedure and primary control of arterial pulsating bleeding or major venous hemorrhage by sutures, ligations, vascular clips, or point electrocautery

Exclusion Criteria:

* Indication for emergency surgery
* Participate in other clinical trials in the past 3 months
* Obvious hematologic disorder (as judged by the investigator from anemia and coagulation dysfunction)
* Patients with brain disease, abnormal judgment or mental disorder that does not cooperate with the researcher
* Patients with asthma or allergies
* Patients with severe cardiac disease, metabolic disease or endocrine disorders
* Immunodeficient patients (AIDS)
* Pregnancy, breastfeeding females
* Skin infection in the field of the targeted incisional area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Hemostatic time | 10 minutes
  Hemostatic time began to calculate when gauze was applied.

SECONDARY OUTCOMES:
Postoperative drainage volume | In the first day after surgery
  Drainage volume through the site
Postoperative drainage time | Up time to removal of wound drain, an expected average of 1 week
  The duration of drainage
Hospital stay | Up time to discharge from hospital,an expected average of 3 weeks
  Total hospital stay
Postoperative hospital stay | Up time to discharge from hospital,an expected average of 2 weeks
  Total postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jialin Zhang, Ph.D/MD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- Hepatobiliary Surgery Department of the First Hosptial of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No